CLINICAL TRIAL: NCT01172665
Title: University of Chicago Celiac Disease Database
Brief Title: Celiac Disease Database
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16103A
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Celiac Disease
Keywords: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The focus of this study is to create a database containing information about patients with celiac disease. This database will allow us to examine clinical and epidemiologic features of the University of Chicago Medical Center patient population. We have the largest population of patients with celiac disease in the mid-West and as such this study using information gathered from our database can greatly contribute to our current understanding of this disease.

DETAILED DESCRIPTION:
This database will allow us to examine clinical and epidemiologic features of the University of Chicago Medical Center patient population.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient at The University of Chicago Medical Center
* Clinical diagnosis of celiac disease or gluten sensitivity

Exclusion Criteria:

* Currently being treated at a healthcare facility other than The University of Chicago Medical Center
* Not diagnosed with celiac disease or gluten sensitivity

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both pediatric and adult patients of The University of Chicago Medical Center who have been diagnosed with celiac disease or gluten sensitivity.
Sampling Method: Non-Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Verma, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States